CLINICAL TRIAL: NCT02805465
Title: Comparison of His Bundle Pacing (HBP) and Bi-Ventricular Pacing(BiVP) in Heart Failure (HF) Patients With Atrial Fibrillation (AF) Who Need Atrial-Ventricular Node (AVN) Ablation
Brief Title: Comparison of His Bundle Pacing and Bi-Ventricular Pacing in Heart Failure With Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: HT-Med Company (Unknown); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Shanghai Zhongshan Hospital (Other); Jiangsu People's Hospital (Unknown); Wuhan Asia Heart Hospital (Other); Sir Run Run Shaw Hospital (Other); Shanxi People's Hospital (Unknown)
Responsible Party: Principal Investigator, Weijiang Huang, Dean of Cardiology, First Affiliated Hospital of Wenzhou Medical University, First Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FirstWenzhouMU001
Record Dates: First submitted 2016-05-30; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Heart Failure; Atrial Fibrillation
Keywords: Heart Failure; Atrial Fibrillation; CRT; BiVP; HBP
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HBP Group (Experimental): CRT Device and His-bundle Pacing. Patients will get His-bundle pacing through a CRT device first for 9 months then switch to Bi-ventricular pacing by the same CRT device for another 9 months.
  Interventions: Device: CRT Device and Bi-ventricular pacing; Device: CRT Device and His-bundle Pacing
- BiVP Group (Active Comparator): CRT Device and Bi-ventricular Pacing. Patients will get BiV pacing for 9 months through a CRT device then switch to His-bundle pacing by the same CRT device for another 9 months.
  Interventions: Device: CRT Device and Bi-ventricular pacing; Device: CRT Device and His-bundle Pacing

INTERVENTIONS:
Device: CRT Device and Bi-ventricular pacing — Bi-ventricular pacing by a CRT device
Device: CRT Device and His-bundle Pacing — His-bundle pacing by a CRT device through the pacing lead at His-bundle region

SUMMARY:
This study is a multicenter, prospective, randomized cross-over study to compare His Bundle Pacing (HBP) with Bi-Ventricular Pacing (BiVP) in HF Patients with AF who need atrial-ventricular node ablation.

DETAILED DESCRIPTION:
Patients who meet the inclusion and exclusion criteria will be enrolled into the study. In the study, both atrial-ventricular node(AVN) ablation and Cardiac Resynchronization Therapy (CRT) implantation are performed with HBP lead implanted and connected with the A port of CRT device. Followed with successful AVN ablation, HBP lead and CRT implantation, patients are 1:1 randomized into BiVP and HBP group for 9 months and then crossover for another 9 months. The primary end points of the study is the change of left ventricular ejection fraction (LVEF) in both HBP and BiV pacing group.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old
* Subject or authorized legal guardian or representative has signed and dated the Informed
* Subject is expected to remain available for follow-up visits at the study center
* Subjects with heart failure NYHA Class II-IV
* Subjects with LVEF no greater than 40%
* Subjects with persistent atrial fibrillation or atrial flutter with uncontrolled ventricular rate

Exclusion Criteria:

* Subjects with the width of ECG Q, R, S wave (QRS) complex >120ms
* Subjects with life expectancy less than 3 years
* Subjects with mechanical right heart valve
* Subjects with primary valvular disease
* Subjects with heart transplant, or is currently on a heart transplant list
* Subjects who are pregnant, or of childbearing potential and not on a reliable form of birth control
* Subjects with significant renal dysfunction, as manifested by serum creatinine level >2.5 mg/dl or ≥275 μmol/L or estimated glomerular filtration rate (GFR) ≤30 mL/min/1.72 m2, which is documented within the 30 days prior to enrollment or at baseline.
* Subjects with significant hepatic dysfunction, as evidenced by a hepatic function panel (serum) > 3 times upper limit of normal, which is documented within the 30 days prior to enrollment or at baseline.
* Subjects with chronic or treatment-resistant severe anemia (hemoglobin <10.0 g/dL), which is documented within the 30 days prior to enrollment or at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Change of LVEF(%) from baseline in HBP and BiV Group | 18 months

SECONDARY OUTCOMES:
Change of 6min walking distance (m) from the baseline | 18 months
Change of LV end diastolic diameter(mm) from baseline | 18 months
Change of LV end systolic diameter(mm) from baseline | 18 months
The number of heart failure hospitalization after the procedure group | 18 months
Change of Quality of Life | 18 months
  The Short Form (36) Health Survey (SF-36) Questionnaire
Change of Average sensing amplitude (V) | 18 months
Change of average pacing threshold (V) | 18 months
Change of average pacing impedance (ohm) | 18 months
Change of New York Heart Association (NYHA) Classification from baseline | 18 months
The number of patients with heart failure hospitalization after the procedure | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Weijian Huang, MD, Principal Investigator — Wenzhou 1st Affliated Hopsital, Wenzhou Medical University
Locations (1):
- First Affliated Hospital, Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang W, Wang S, Su L, Fu G, Su Y, Chen K, Zou J, Han H, Wu S, Sheng X, Chen X, Fan X, Xu L, Zhou X, Mao G, Ellenbogen KA, Whinnett ZI. His-bundle pacing vs biventricular pacing following atrioventricular nodal ablation in patients with atrial fibrillation and reduced ejection fraction: A multicenter, randomized, crossover study-The ALTERNATIVE-AF trial. Heart Rhythm. 2022 Dec;19(12):1948-1955. doi: 10.1016/j.hrthm.2022.07.009. Epub 2022 Jul 14. PMID 35843465